CLINICAL TRIAL: NCT02879344
Title: Extra Corporeal Membrane Oxygenation in the Acute Respiratory Distress Syndrome: Utility of a Biomarker to Assess the Membrane Efficiency in Improving Oxygenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-17; 2012-A00677-36 (Other: ANSM)
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2016-08

CONDITIONS: Extra Corporel Membrane Oxygenation and Mciroparticles
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patient undergoing ECMO (Other)
  Interventions: Other: Blood draw

INTERVENTIONS:
Other: Blood draw

SUMMARY:
ECMO (extra-corporeal membrane oxygenation) is a blood oxygenation technical and purification of carbon dioxide by means of an extracorporeal circulation using a pump (identical to those used in cardiac surgery) and a membrane permitting gas exchange. This technique is used for almost 40 years in the acute respiratory distress syndrome (ARDS) but benefited from many technology improvements over the past 10 years.

The circuit is now fully pre-heparin, not imposing obtaining activated partial thromboplastin time (aPTT) high. Centrifugal pumps limit the risk of intravascular hemolysis. The multi-perforated drainage cannula in place in femoral vein or jugular no longer need to maintain hypervolaemia to ensure sufficient flow.

The membrane ensuring gas exchange is now polymethylpentene. This hollow fiber system ensures the gas exchange.

In light of recent technical improvements, manufacturers indicate that the membranes can be used for 3 weeks. However, after a few days of use, fibrinoplaquettaires microthrombi form at the ECMO circuit, up from cannulas up to the oxygenator, decreasing membrane efficiency and imposing more early changes of the circuit. This hypercoagulable state was revealed through the study of classical plasma markers of coagulation. There is not so far from reliable predictive marker of thrombus formation, indicating a need to change the circuit.

The production of microparticles (MPs) is a characteristic of cells subjected to an activation or apoptosis. MPs are membrane Smaller fragments released into the extracellular milieu after rupture of the asymmetry of the distribution of membrane phospholipids and characterized by the presence of phosphatidylserine (PhtdSer) on their surface, as well as various antigens expressed by their cells of origin. The PhtdSer is a pro-coagulating surface on which are going to assemble the enzymes responsible for the formation of thrombin and increases proportionally the TF activity ultimately leading to fibrin polymerization in the vessels.

The vesiculation phenomenon exists in healthy subjects. In human pathology, many examples emphasize the fundamental role of MP in clotting or thrombosis. The PM generating fault is associated with bleeding disorders (Scott syndrome, dysvésiculation syndrome). Conversely, high circulating levels of MP are found in many thrombotic diseases (myocardial infarction, diabetes, antiphospholipid antibody syndrome, preeclampsia ...). Platelet and intense monocyte endothelial activation, observed in sepsis and severe trauma, is accompanied by the generation of procoagulant MP carriers of tissue factor (TF). These MP diffuse into the vascular compartment pathogenic potential may exacerbate inflammatory and thrombotic responses and play a leading role in triggering the DIC.

More recently, various studies have shown that the microparticles are not only activation markers or injury, but also cellular elements having a true pathogenic role. Because they contain or express on their surface various biological effector (adhesion molecules, tissue factor, inflammatory mediators or apoptogenic, growth factor ...) the microparticles are able to interact with their environment and modulate cellular very different way the properties of target cells. And platelet or leukocyte microparticles could actively participate in the thrombotic process by increasing adhesion of monocytes and endothelial cells, or by inducing endothelial procoagulant response.

ELIGIBILITY:
Inclusion Criteria:

* Pateint undergoing ECMO and invasive ventilation with PaO2/FiO2 < 70 mmHg

Exclusion Criteria:

* BMI > 0.75 kg.cm-1
* Advanced multi-visceral failure scored with SOFA>17 for ARDS patient<7 days or SOFA > 11 for ARDS patient>7 days .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Assesement of microparticles percentage produced in patient undergoing ECMO | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Christophe GUERVILLY, MD, Principal Investigator — Assistance Publique Hopitaux De Marseille; Urielle DESALBRES, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No